CLINICAL TRIAL: NCT01257893
Title: Aspirin Resistance in Women With Migraine
Acronym: ARWM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Swedish Medical Center (Other)
Collaborators: University of Washington (Other); National Headache Foundation (Unknown); Wadsworth Foundation (Unknown); Accumetrics, Inc. (Industry)
Responsible Party: Jill T. Jesurum, Ph.D., Scientific Director, Swedish Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: 4959S-10
Record Dates: First submitted 2010-12-08; First posted 2010-12-10 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Episodic Migraine; Chronic Migraine
Keywords: migraine; chronic migraine; migraine with aura; migraine without aura; aspirin; platelets
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Migraine without Aura | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspirin 81 mg (Experimental): Subjects will take 81 mg aspirin per day for 10-14 consecutive days
  Interventions: Drug: Aspirin (acetylsalicylic acid)
- Placebo (Placebo Comparator): Subjects will take matching placebo capsule (excipient: methylcellulose) for 10-14 consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin (acetylsalicylic acid) — Aspirin one 81 mg capsule per day for 10-14 consecutive days
  Arms: Aspirin 81 mg
Drug: Placebo — 1 placebo capsule identical in appearance and excipient to aspirin capsule per day for 10-14 consecutive days
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the rates of aspirin resistance (high residual platelet reactivity) between women with episodic and chronic migraine and women without migraine.

Emerging evidence suggests that migraineurs, especially women < 45 years who have aura, have an increased risk of stroke and myocardial infarction (MI, or heart attack). The mechanism linking migraine, stroke and MI is unclear although increased platelet activation and aggregation observed during and between migraine attacks may be a plausible theory.

Aspirin is an inexpensive, relatively safe antiplatelet drug that reduces the risk of stroke and MI. Preliminary data suggest that aspirin's (325mg) therapeutic effect on platelet inhibition may be reduced in migraineurs (i.e., aspirin resistance), thus limiting aspirin's effectiveness at preventing stroke and MI risks in persons with migraine. Additional research is warranted to confirm these findings in migraineurs because daily, low-dose aspirin 81 mg is the recommended first line therapy for primary and secondary prevention of stroke and MI

The researchers hypothesize that resistance to aspirin 81mg may occur more frequently in women with episodic and chronic migraine than in women without migraine. The findings may have important implications for women who have migraine and use aspirin to prevent migraine symptoms or comorbidities associated with migraine including stroke and MI.

DETAILED DESCRIPTION:
To test the hypothesis that the rate of aspirin resistance is greater in women with episodic and chronic migraine than in women without migraine, a three-group, randomized, double-blind, placebo-controlled, crossover design will be used to test the effects of aspirin 81 mg on platelet reactivity. Subjects will be randomized to treatment order (A) aspirin 81 mg for 10-14 consecutive days followed by placebo for 10-14 consecutive days or (B) placebo for 10-14 consecutive days followed by aspirin 81 mg for 10-14 consecutive days. Other than treatment order, subjects will be treated equally. Study procedures will be performed at the University of Washington, and the duration of the study per subject will be approximately 28 days. Endpoints include: a) Aspirin Reaction Units (ARU) using a point-of-care assay (VerifyNow Aspirin™; Accumetrics, San Diego, CA); b) serum thromboxane B2; and c) percent platelet inhibition on aspirin. Assessment of adherence to study regimen will be assessed by serum salicylate, medication diaries, and pill counts. Data will also be collected on migraine frequency, burden, disability, and medications used to treat headache. Subjects will maintain a migraine diary for the duration of the study (28 days). The target sample will include women with episodic migraine (n=40; n=20 MA, n=20 MO), women with chronic migraine (n=40) and non-migraine controls (n=40).

The specific aims of the study are as follows:

* Compare the rate of aspirin resistance between women with and without migraine following 10-14 consecutive days of aspirin 81 mg treatment
* Compare the rate of aspirin resistance between women who have episodic migraine and chronic migraine following 10-14 consecutive days of aspirin 81 mg treatment
* Compare the rate of aspirin resistance between women who have migraine with aura (MA) and migraine without aura (MO) following 10-14 consecutive days of aspirin 81 mg or placebo treatment
* Compare the rate of aspirin resistance between women who have migraine with high monthly migraine frequency and low monthly migraine frequency following 10-14 consecutive days of aspirin 81 mg treatment

ELIGIBILITY:
Inclusion Criteria:

* Women 18-50 years of age, of childbearing potential
* Able to read, speak, and understand English -- except if patient is blind, in which case only the ability to understand English is required.

Episodic Migraine Group:

* Documented diagnosis of episodic migraine for a 2-year period preceding enrollment, using the International Headache Society (IHS) criteria.
* Frequency of 2-14 migraine days in the three months prior to enrollment.
* Equal numbers (n=20 each) will have a documented diagnosis of migraine with aura (MA) and migraine without aura (MO).
* For women who have a diagnosis of MA, focal neurologic symptoms must precede or accompany the headache (aura) for at least one headache in the 12 months prior to enrollment.

Chronic Migraine Group:

* Frequency of ≥ 15 headache days per month for ≥ 3 months.
* On at least 8 days per month for ≥ 3 months headache has fulfilled criteria for pain and associated symptoms of MO.

Control group:

- No diagnosis of migraine, confirmed by the Migraine Assessment Tool.

Exclusion Criteria:

* Pregnancy or lactation
* Post-menopausal, either natural or surgical (bilateral oophorectomy)
* Current prescribed daily medication regimen includes any of the following: warfarin, glycoprotein IIb/IIIa inhibitors (abciximab, tirofiban), antiplatelet agents (clopidogrel, ticlopidine, dipyridamole), or non-steroidal anti-inflammatory drugs (e.g., ibuprofen, naproxen, celecoxib), Vitamin E in doses > 800 IU per day, Omega-3 fatty acids in doses > 3 g/day, willow bark (any amount), aspirin or aspirin-containing medications.
* Aspirin intolerance or allergy, or peptic ulcer disease.
* Platelet count <150,000/µl or >450,000/µl.
* Hemoglobin <10 g/dL.
* History or current diagnosis of myocardial infarction, stroke, coronary artery disease, peripheral arterial disease, diabetes mellitus, or renal disease.
* Unable to tolerate washout of protocol-restricted medications and/or supplements (see #3).
* Family (first-degree relative) or patient history of bleeding or hemorrhagic disorders including von Willebrand Factor Deficiency, Glanzmann Thrombasthenia, Bernard-Soulier Syndrome or myeloproliferative syndromes.
* Major surgical procedure, trauma, blood donation, or major blood loss (>300 cc) within 30 days prior to enrollment.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Aspirin Reaction Units (ARU) | 10-14 days
  Measurement of ARU, indicative of platelet inhibition, using the VerifyNow Aspirin Assay (Accumetrics, San Diego, CA)

SECONDARY OUTCOMES:
Serum thromboxane B2 | 10-14 days
  Aspirin acts by inhibiting production of thromboxane A2 by platelets. Thromboxane B2 is the stable product of thromboxane A2.

CONTACTS AND LOCATIONS:
Overall Officials: Jill T. Jesurum, Ph.D., Principal Investigator — Swedish Medical Center; Cindy J. Fuller, Ph.D., Study Director — Swedish Medical Center; Sylvia M. Lucas, MD, PhD, Study Chair — University of Washington; Natalia Murinova, MD, Study Chair — University of Washington
Locations (1):
- The University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Jesurum, J.T., Fuller, C.J., Lucas, S.M., Murinova, N., Truva, C.M., McGee, E.A., Reisman, M. High prevalence of aspirin resistance in migraineurs. Cephalalgia 2009; 29 (Suppl. 1): 138.
- [Background] Jesurum, J.T., Fuller, C.J., Lucas, S.M., Murinova, N., Hales, L.E., McGee, E.A. The association between migraine frequency and platelet activation in episodic migraine: a pilot study. Cephalalgia 2009; 29 (Suppl. 1); 2009.